CLINICAL TRIAL: NCT07117734
Title: Evaluating the Suitability of YouTube as a Platform for Enhancing Dynamic Balance
Brief Title: Reliability and Quality of YouTube Videos Related to Balance Exercise
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Ali Zorlular, Assistant Professor, Nigde Omer Halisdemir University
Other Study IDs: Balance and Youtube
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Dynamic Balance; Balance
Keywords: balance; video; youtube

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: An Evaluation of the Quality and Informational Content of Balance Exercise Training Videos Published on YouTube. — In the study, there will be no participant groups; YouTube videos searched using the keyword "balance exercise" will be evaluated based on specific criteria.

SUMMARY:
This study aimed to find out how useful and trustworthy YouTube videos are when it comes to teaching dynamic balance exercises. Researchers watched and analyzed selected videos to check the accuracy of the information, how reliable the sources were, and how well the videos were made to help viewers learn. The goal was to help people find better-quality videos for safe and effective balance training.

ELIGIBILITY:
Inclusion Criteria:

* Videos retrieved using the keyword "dynamic balance exercise"
* Videos in English
* Presence of audio narration or explanation
* Demonstration of exercise practices within the video content

Exclusion Criteria:

* Duplicate videos (i.e., videos with identical or highly similar content)
* Videos with unclear or unintelligible audio and/or visual content

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Videos searched on the YouTube platform using the keyword "balance exercises."
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Quality of videos | From registration until the end of the second week
  The DISCERN tool is a standardized questionnaire developed to enable researchers to systematically evaluate the quality of health information related to treatment options. The instrument comprises 15 specific items followed by an overall assessment question aimed at rating the general quality of the information provided

SECONDARY OUTCOMES:
Quality of videos 2 | From registration until the end of the second week
  The overall quality of each video was evaluated using the 5-point Global Quality Scale (GQS), a widely used instrument for assessing the comprehensiveness and clarity of health information. According to the rating criteria, videos receiving a score of 1 or 2 were classified as low quality, a score of 3 as moderate quality, and scores of 4 or 5 as indicative of high quality.

OTHER OUTCOMES:
Video popularity | From registration until the end of the second week
  Video popularity was quantitatively assessed using two validated metrics: the Video Power Index (VPI), calculated as the ratio of likes to the total number of likes and dislikes multiplied by 100 (likes/(likes+dislikes))×100 and the View Ratio (VR), defined as the number of views divided by the number of days since the video was uploaded (views/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Bor Faculty of Health Sciences, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Erdem MN, Karaca S. Evaluating the Accuracy and Quality of the Information in Kyphosis Videos Shared on YouTube. Spine (Phila Pa 1976). 2018 Nov 15;43(22):E1334-E1339. doi: 10.1097/BRS.0000000000002691. PMID 29664816
- [Result] Anastasio AT, Tabarestani TQ, Bagheri K, Bethell MA, Prado I, Taylor JR, Adams SB. A New Trend in Social Media and Medicine: The Poor Quality of Videos Related to Ankle Sprain Exercises on TikTok. Foot Ankle Orthop. 2023 May 4;8(2):24730114231171117. doi: 10.1177/24730114231171117. eCollection 2023 Apr. PMID 37151477
- [Result] Sari F, Bazancir Apaydin Z, Sari S. Assessment of reliability and quality of YouTube(R) exercise videos in people with rheumatoid arthritis. Physiother Theory Pract. 2025 Feb;41(2):362-369. doi: 10.1080/09593985.2024.2334753. Epub 2024 Mar 27. PMID 38536002
- [Derived] Zorlular A, Zorlular R. Evaluating online video platforms for dynamic balance exercises: a focus on YouTube. Phys Sportsmed. 2025 Dec 1:1-8. doi: 10.1080/00913847.2025.2597183. Online ahead of print. PMID 41307528